CLINICAL TRIAL: NCT07140393
Title: An Open, Multicenter Phase IB/II Clinical Study of HRS-4508 in Combination With Other Anti-tumor Therapy for Solid Tumor
Brief Title: A Study of HRS-4508 in Combination With Other Anti-tumor Therapy for Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4508-202-BC
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HRS-4508+ Capecitabine (Experimental)
  Interventions: Drug: HRS-4508+ Capecitabine
- HRS-4508+ Trastuzumab (Experimental)
  Interventions: Drug: HRS-4508+ Trastuzumab
- HRS-4508+ Trastuzumab+ Pertuzumab (Experimental)
  Interventions: Drug: HRS-4508+ Trastuzumab+ Pertuzumab
- HRS-4508+ Trastuzumab+ Capecitabine (Experimental)
  Interventions: Drug: HRS-4508+ Trastuzumab+ Capecitabine
- Trastuzumab+ Capecitabine (Experimental)
  Interventions: Drug: Trastuzumab+ Capecitabine
- HRS-4508+A1811 (Experimental)
  Interventions: Drug: HRS-4508+A1811

INTERVENTIONS:
Drug: HRS-4508+ Capecitabine — HRS-4508+ Capecitabine
  Arms: HRS-4508+ Capecitabine
Drug: HRS-4508+ Trastuzumab — HRS-4508+ Trastuzumab
  Arms: HRS-4508+ Trastuzumab
Drug: HRS-4508+ Trastuzumab+ Pertuzumab — HRS-4508+ Trastuzumab+ Pertuzumab
  Arms: HRS-4508+ Trastuzumab+ Pertuzumab
Drug: HRS-4508+ Trastuzumab+ Capecitabine — HRS-4508+ Trastuzumab+ Capecitabine
  Arms: HRS-4508+ Trastuzumab+ Capecitabine
Drug: Trastuzumab+ Capecitabine — Trastuzumab+ Capecitabine
  Arms: Trastuzumab+ Capecitabine
Drug: HRS-4508+A1811 — HRS-4508+A1811
  Arms: HRS-4508+A1811

SUMMARY:
The study is being conducted to evaluate the efficacy, safety, and ORR of HRS-4508 combination with other anti tumor therapy in subjects with solid tumor ; to evaluate HRS4508 DLT, MTD and RP2D, to evaluate the incidence and severity of adverse events (AE)/serious adverse events (SAE) (rated based on CTCAE v5.0), to evaluate ORR by researchers based on RECIST v1.1, to evaluate the pharmacokinetic (PK) characteristics of HRS-4508 SHR-1811, Capecitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old; Both men and women are welcome;
2. The mixed cell types need to be confirmed by histology or cytology, and the dominant cell morphology, unresectable or metastatic .
3. ECOG ratings of 0 or 1.
4. Expected survival period ≥ 12 weeks.
5. At least one measurable lesion outside the central nervous system that meets the RECIST v1.1 standard definition.
6. Willing to participate and comply with the requirements of the research protocol, and willing to cooperate with follow-up visits.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis. Subjects with a history of meningeal metastasis or current meningeal metastasis
2. There have been significant severe infections and major surgeries in the past 4 weeks
3. Existence of previous or concurrent malignant tumors
4. Difficult to treat nausea, vomiting, or other gastrointestinal diseases that affect the use of oral medication
5. Having undergone major surgeries other than diagnosis or biopsy within 28 days prior to the first administration;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
HRS4508 DLT | 3 weeks
HRS4508 MTD | 12 weeks
HRS4508 RP2D | 12 weeks
The incidence and severity of adverse events (AE)/serious adverse events (SAE) (rated based on CTCAE v5.0) | 2 years
Objective response rate (ORR) | 1 year

SECONDARY OUTCOMES:
Blood concentrations of HRS-4508 | 15 weeks
Blood concentrations of SHR-A1811 | 9 weeks
Blood concentrations of Capecitabine | 2 weeks
Objective response rate (ORR) | 1 year
Best overall efficacy (BOR) | 1 year
Duration of response (DoR) | 1 year
Progression free survival (PFS) | 1 year
Disease control rate (DCR) | 1 year
Overall survival (OS) | 2 year
The incidence and severity of adverse events (AE)/serious adverse events (SAE) (rated based on CTCAE v5.0) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided